CLINICAL TRIAL: NCT03689270
Title: Central Corneal Thickness Assessment After Phacoemulsification: Subluxation Versus Divide-and-Conquer
Brief Title: Corneal Edema After Phacoemulsification
Acronym: COPHA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-12Obs-CHMRT
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Cataract
Keywords: subluxation; Divide and conquer
MeSH Terms: conditions — Cataract; Joint Dislocations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subluxation: Nucleus is hydrodissected until it lilts above the capsular bag, rotated to face the incision then tumbled and emulsification continues from the opposite equator outside in until complete
  Interventions: Procedure: Subluxation
- Divide and Conquer: Cataract nucleus is fragmented into 4 pieces then aspirated by ultrasonic vibration
  Interventions: Procedure: Divide and conquer

INTERVENTIONS:
Procedure: Subluxation — One pole of The nucleus is hydrodissected until it lilts above the capsular bag. The tilted nucleus is rotated to face the incision and remaining half nucleus is then tumbled and emulsification continues from the opposite equator outside in until complete.
  Groups: Subluxation
Procedure: Divide and conquer — Cataract nucleus is fragmented into 4 pieces then aspirated by ultrasonic vibration
  Groups: Divide and Conquer

SUMMARY:
To compare the impact of two phacoemulsification techniques (subluxation versus divide-and-conquer) on postoperative corneal edema at postoperative hour 1 and day 4.

DETAILED DESCRIPTION:
Phacoemulsification is the procedure of choice for most surgeons performing cataract surgery. Alternative techniques have been in development over the last twenty years, with the hope of optimizing operating times, total ultrasound energy used, patient safety, patient satisfaction and visual recovery associated with cataract surgery.

Divide-and conquer is the parent nucleofracture technique.The subluxation technique is a newer technique that is less frequently used because of an increased risk of corneal endothelium damage.

The aim of this comparative study was to evaluate corneal edema immediately after surgery performed with the subluxation technique versus divide-and-conquer. Corneal edema was determined by measuring central corneal thickness (CCT).

ELIGIBILITY:
Inclusion Criteria:

* The presence of a senile cataract with equivalent grades and history of visual acuity regression
* Informed written consent

Exclusion Criteria:

* Patients with total white cataract
* With history of ocular surgery and other eye diseases (corneal pathology, uveitis, glaucoma)
* With systemic diseases with the potential to affect vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent phacoemulsification cataract surgery over a 6-month period.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Corneal edema preoperative | Day 1
  Central corneal thickness measurements were taken preoperatively

SECONDARY OUTCOMES:
Corneal edema postoperative | Day 4
  Central corneal thickness measurements were taken postoperative day 4